CLINICAL TRIAL: NCT03196167
Title: Efficacy and Safety of Sugammadex (2mg/kg) to Shorten Time-to-extubation Among Postoperative ICU Patients Following AVR, CABG Surgery, or AVR/CABG Surgery- a Prospective Randomized Placebo-controlled Trial.
Brief Title: Sugammadex and Decreased Time to Extubation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2000021124
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Results first posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Coronary Artery Bypass Graft and/or Aortic Valve Replacement Surgery
Keywords: sugammadex; extubation; CABG, AVR, CABG/AVR combination
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Intervention Model Description: Patients will be enrolled using 1:1 randomization between active ingredient (intervention) and control arms, to be assigned randomly using a computer generated algorithm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The administration of the study and placebo compounds will be performed by CTICU nurses who will receive the drugs in a blinded fashion from the departmental research pharmacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sugammadex (Experimental): Research pharmacy will provide the Sugammadex (2m/kg) vs. Placebo in a syringe.
  Interventions: Drug: Sugammadex
- Placebo (Placebo Comparator): Research pharmacy will provide the Sugammadex (2m/kg) vs. Placebo in a syringe.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sugammadex — The administration of the study and placebo compounds will be performed by CTICU nurses who will receive the drugs in a blinded fashion from the departmental research pharmacy.
  Other Names: Bridion
  Arms: Sugammadex
Other: Placebo — The administration of the study and placebo compounds will be performed by CTICU nurses who will receive the drugs in a blinded fashion from the departmental research pharmacy.
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate faster time to extubation after arrival in the cardiothoracic intensive care unit (ICU) in patients undergoing isolated coronary artery bypass grafting (CABG), AVR and AVR/CABG combination who receive Sugammadex as compared to placebo.

DETAILED DESCRIPTION:
Primary Efficacy Objective: To demonstrate faster time to extubation after arrival in the cardiothoracic ICU in patients having a CABG who receive Sugammadex 2mg/kg as compared to placebo.

Hypotheses: We hypothesize that the use of Sugammadex for reversal of residual neuromuscular blockade in adults undergoing CABG, AVR or CABG/AVR combination surgery in the cardiothoracic ICU will significantly decrease the time to extubation.

Prolonged intubation after cardiac surgery continues to be a common clinical challenge and is associated with significant risks and costs(1-5). Despite a Class I recommendation by the American College of Cardiology supporting care directed towards early postoperative extubation after low to medium risk Coronary Artery Bypass Grafting (CABG) surgeries (6), a sizable proportion of patients continue to have a prolonged course of cardiothoracic intensive care unit (CTICU) intubation(1). Residual neuromuscular blockade (NMB) continues to be one of the key factors leading to prolonged intubation after cardiac surgery(7). It is also a significant contributor to postoperative pulmonary and respiratory complications including hypoxia, upper airway obstruction; and decreased oxygen saturation - often prompting reintubation in critical care units(8-10). Due to the profound effects that neuromuscular reversal agents other than Sugammadex have when used in combination with muscarinic acetylcholine receptor antagonists on the autonomic nervous system and patient hemodynamics, these traditional reversal drugs are rarely used in the postoperative cardiac surgery patient population (11) as opposed to other general surgical cases.

Sugammadex, a gamma-cyclodextrin drug, rapidly reverses neuromuscular blockade by encapsulating the non-depolarizing amino steroids agents(12) and is not associated with cardiovascular effects that are commonly seen with traditional NMB reversal agents(13). It can also reverse NMB more quickly and predictably than existing agents(14). However, there have been sporadic reports of hypotension(15), anaphylaxis(16), elongated a PTT(17) with the use of Sugammadex. Additionally, although the FDA currently lists Sugammadex as indicated for reversal of neuromuscular blockade induced by rocuronium and vecuronium in adults undergoing surgery,(18) its use in the post cardiac surgery setting is limited due to lack of supportive data. In this context, the present study aims to test the effectiveness of a pragmatic and broadly applicable care pathway for shortening time to extubation among patients in the cardiothoracic ICU who have undergone isolated CABG, AVR or CABG/AVR combination procedure. The FDA-approved package insert is attached as an appendix to this application.

Study design: Prospective, randomized, double blind, single center placebo-controlled trial.

Number of participants: 110 enrolled with assumed randomization of 90 using 1:1 randomization between active ingredient (intervention) and control arms, to be assigned randomly using a computer generated algorithm.

Subject Recruitment: Subjects will be consented in the collaborating surgeons offices or in pre-admission testing. Every effort will be made to consent subjects prior to day of surgery. If a patient is referred or identified any time after those visits, they may be consented in the preoperative area.

Anesthetic management per protocol:For enrolled patients, anesthetic management will be left to the discretion of the attending anesthesiology provider. As per our usual clinical practice, Rocuronium or vecuronium will be used as the non-depolarizing NMB and that where sedation is desired and appropriate, The patients will be transferred to the CTICU intubated and on a propofol infusion and/or dexmedetomidine per our usual clinical practice.

Upon CTICU arrival, determination of continued eligibility will be determined. If the decision is made to continue on a fast-track extubation pathway, eligible patients will be randomized, investigational pharmacy will be contacted for study drug. 30 minutes after the ICU admission, propofol will be discontinued. Precedex may be continued per clinical discretion. The participant will be randomized to either receive Sugammadex or placebo. A qualitative train-of-four measurement will be obtained. The administration of the study and placebo compounds will be performed by CTICU nurses who will receive the drugs in a blinded fashion from the departmental research pharmacy. The level of neuromuscular blockade will be measured by accelerometer before and after the drug/placebo administration by the research coordinator. This will be done by placing a sheet over the limb being tested, so that the clinical team remains blinded to the results of the drug /placebo administration. The study drug will be supplied by Merck. Patients will be initiated on SIMV with 40% FiO2, tidal volumes 8-10 ml/kg and PEEP of 5.

Ten minutes after the drug administration, if the patient is able to lift head and remains hemodynamically stable, the patient will be switched to CPAP mode of ventilation for 30 minutes. At the end of the CPAP trial tidal volumes, Rapid Shallow Breathing Index (RSBI) and ABG will be assessed. The patient will be extubated if he/she is not hypoxic/ hypercarbic, has RSBI<100 and has TV >300 cc. The final clinical decision to extubate the patients will be taken by the CTICU team.

If a patient fails the 30 minute CPAP criteria, the ICU intensivist will be immediately notified. Every attempt will be made to correct the underlying cause of CPAP failure, and a prompt reassessment will be made as deemed appropriate by the intensivist to reattempt CPAP versus continuing controlled mechanical ventilation.

It is estimated conservatively that the study personnel will randomize 3 patients per week allowing for data collection to be completed within 1 year of study commencement. Data analysis and dissemination of findings will be conducted over the subsequent 6 months by the study institution investigators per the publication plan below.

Blinded analyses of the data will be performed by the study investigators along with the departmental statistician in the Department of Anesthesiology at the Yale School of Medicine.

Variables/Time Points of Interest: The primary outcome is the time to extubation, which will be the duration from arrival to the ICU to the extubation time. Participants' blood pressure, heart rate, and chest tube output will be tracked from arrival to the CTICU until extubation per ICU protocol.

Statistical Methods:Baseline comparability. We expect that the randomization process will produce reasonably comparable groups. However, the adequacy of the randomization will be assessed by comparing the distribution of baseline demographic and clinical characteristics among the intervention groups. Comparability for continuous variables will be examined graphically and by summary statistics (means, medians, quartiles, etc.). Categorical variables will be examined by calculating frequency distributions.

Proposed statistical test/analysis: Positively skewed variables will be log-transformed prior to hypothesis testing. For the primary outcome, a two-sided Student's t-test will be used to compare the time to extubation between the two groups. If necessary, covariate adjustment will be made using the multiple linear regression analysis method. Differences between means and 95% confidence intervals will be estimated to describe the magnitude of intervention difference between the two groups. As part of sensitivity analyses, the time-to-extubation outcome will be also analyzed by the Cox regression model. To compare the categorical adverse events between two groups, chi-square test or Fisher's exact test will be used.

Missing Data: Prevention is the most obvious and effective manner to control bias and loss of power from missing data. Therefore, several strategies (e.g., timely data entry and daily missing data report) will be imposed to limit the likelihood that missing data will occur during this study. This protocol will follow the intention to treat principle, requiring follow-up of all subjects randomized regardless of the actual treatment received.

Power analysis: Our 'in-house' historical data (n = 73) showed that after excluding outliers greater than the 80th percentile, patients undergoing isolated CABG demonstrated a mean of 8.39 hours to extubation (SD 2.89). Although we anticipate a Hawthorne effect demonstrating reduced time to extubation in both the active and placebo arms of the present study, we have conservatively chosen to maintain power based on historical data. We therefore estimate that 45 subjects per group will give us 90% power to detect a clinically relevant effect size of 2-hours difference between active and placebo groups at an alpha value of 0.05 using a two-sided two-sample t-test. To allow for post consent, pre-randomization study drop out, we will aim to enroll a total of 110 (90 + 20 = 110) subjects.

Per-protocol Sensitivity Analysis: In parallel with the primary analysis, if exclusions above occur post randomization but prior to drug administration, the investigators will conduct a parallel "per-protocol" sensitivity analysis.

Drug supplies will be supplied by the sponsor.

Adverse Experience Reporting: Throughout the duration of the study, researchers will adhere to good clinical practice and the guidelines of the institution. Patient vitals will be continuously monitored during and after the administration of the test drug. A data and safety monitoring board (DSMB) consisting of the head nurse and a senior critical care staff will meet monthly to discuss any serious events. Any incidence of anaphylaxis or unexplained hypotension requiring initiation of pressors or cardiac pacing within 5 minutes of drug administration will be reported an evaluated. Increases in chest tube output considered clinically significant by the critical care team will be noted. Any of these adverse events will trigger an analysis by the DSMB. If the DSMB determines that study drug may be causing an increase in adverse events, the study will be suspended until the DSMB is able to fully review the events and make a recommendation in consultation with the Yale Human Investigations Committee. The local Merck research representative will also be notified about the events. If the data monitoring board and/or institutional review board (IRB) view that the study is unsafe, the study will be discontinued.

Specific Safety Events to Be Reported During Manuscript Preparation: For manuscript preparation, the rates of hypotension, anaphylaxis, and bleeding (i.e. Chest Tube output) will be reported and compared between active and placebo groups.

ELIGIBILITY:
Inclusion Criteria:

* All elective ARV, CABG cases, on-pump or off-pump, and CABG/AVR in adult patients with preoperative left ventricular ejection fraction (LVEF) ≥45%.

Exclusion Criteria:

* Emergency/unplanned cases.
* EF<45% or moderate /severe RV dysfunction.
* Estimated GFR < 30 mL/min.
* Patients on supplemental oxygen at baseline (home oxygen).
* BMI>40 (calculated as the patient's weight in kilograms divided by the square of the patient's height in meters).
* Patients with chronic opioid use preoperatively.
* Patients with known neuromuscular disorders preoperatively.
* Patients with a known sensitivity to Rocuronium or to Sugammadex.
* Patients with known cognitive deficits preoperatively.

Exclusions after recruitment but prior to randomization:

* Postoperative Bleeding (chest tube output >100cc/hr ).
* Treatment of anaphylactoid reaction intraoperatively.
* Patient's temperature<35.5 or >38.3 degree Celsius at the time of ICU arrival.
* Determination that the patient will require prolonged mechanical ventilation possibly requiring muscle relaxation based on the intraoperative course and clinical judgment of the study PI or collaborating intensivists.
* Intraoperative hypoxia or on arrival to the ICU. (Please see Study Flowchart).
* Cardiac arrest.
* Sudden arrhythmia (Ventricular tachycardia runs/sudden bradycardia with improper pacemaker detection/function) precluding fast-track extubation protocol.
* Need for inotrope initiation precluding fast-track protocol.
* Postoperative ST changes.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-05-13 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Bardia, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hefner JL, Tripathi RS, Abel EE, Farneman M, Galloway J, Moffatt-Bruce SD. Quality Improvement Intervention to Decrease Prolonged Mechanical Ventilation After Coronary Artery Bypass Surgery. Am J Crit Care. 2016 Sep;25(5):423-30. doi: 10.4037/ajcc2016165. PMID 27587423
- [Background] Cislaghi F, Condemi AM, Corona A. Predictors of prolonged mechanical ventilation in a cohort of 5123 cardiac surgical patients. Eur J Anaesthesiol. 2009 May;26(5):396-403. doi: 10.1097/EJA.0b013e3283232c69. PMID 19276979
- [Background] Myles PS, Daly DJ, Djaiani G, Lee A, Cheng DC. A systematic review of the safety and effectiveness of fast-track cardiac anesthesia. Anesthesiology. 2003 Oct;99(4):982-7. doi: 10.1097/00000542-200310000-00035. No abstract available. PMID 14508335
- [Background] Hawkes CA, Dhileepan S, Foxcroft D. Early extubation for adult cardiac surgical patients. Cochrane Database Syst Rev. 2003;(4):CD003587. doi: 10.1002/14651858.CD003587. PMID 14583985
- [Background] van Mastrigt GA, Maessen JG, Heijmans J, Severens JL, Prins MH. Does fast-track treatment lead to a decrease of intensive care unit and hospital length of stay in coronary artery bypass patients? A meta-regression of randomized clinical trials. Crit Care Med. 2006 Jun;34(6):1624-34. doi: 10.1097/01.CCM.0000217963.87227.7B. PMID 16614584
- [Background] Hillis LD, Smith PK, Anderson JL, Bittl JA, Bridges CR, Byrne JG, Cigarroa JE, Disesa VJ, Hiratzka LF, Hutter AM Jr, Jessen ME, Keeley EC, Lahey SJ, Lange RA, London MJ, Mack MJ, Patel MR, Puskas JD, Sabik JF, Selnes O, Shahian DM, Trost JC, Winniford MD. 2011 ACCF/AHA Guideline for Coronary Artery Bypass Graft Surgery: executive summary: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Circulation. 2011 Dec 6;124(23):2610-42. doi: 10.1161/CIR.0b013e31823b5fee. Epub 2011 Nov 7. No abstract available. PMID 22064600
- [Background] Hemmerling TM, Russo G, Bracco D. Neuromuscular blockade in cardiac surgery: an update for clinicians. Ann Card Anaesth. 2008 Jul-Dec;11(2):80-90. doi: 10.4103/0971-9784.41575. PMID 18603747
- [Background] Abad-Gurumeta A, Ripolles-Melchor J, Casans-Frances R, Espinosa A, Martinez-Hurtado E, Fernandez-Perez C, Ramirez JM, Lopez-Timoneda F, Calvo-Vecino JM; Evidence Anaesthesia Review Group. A systematic review of sugammadex vs neostigmine for reversal of neuromuscular blockade. Anaesthesia. 2015 Dec;70(12):1441-52. doi: 10.1111/anae.13277. PMID 26558858
- [Background] Murphy GS, Szokol JW, Marymont JH, Greenberg SB, Avram MJ, Vender JS. Residual neuromuscular blockade and critical respiratory events in the postanesthesia care unit. Anesth Analg. 2008 Jul;107(1):130-7. doi: 10.1213/ane.0b013e31816d1268. PMID 18635478
- [Background] Fuchs-Buder T, Nemes R, Schmartz D. Residual neuromuscular blockade: management and impact on postoperative pulmonary outcome. Curr Opin Anaesthesiol. 2016 Dec;29(6):662-667. doi: 10.1097/ACO.0000000000000395. PMID 27755128
- [Background] Murphy GS, Szokol JW, Vender JS, Marymont JH, Avram MJ. The use of neuromuscular blocking drugs in adult cardiac surgery: results of a national postal survey. Anesth Analg. 2002 Dec;95(6):1534-9, table of contents. doi: 10.1097/00000539-200212000-00012. PMID 12456412
- [Background] Welliver M. New drug sugammadex: a selective relaxant binding agent. AANA J. 2006 Oct;74(5):357-63. PMID 17048555
- [Background] Nicholson WT, Sprung J, Jankowski CJ. Sugammadex: a novel agent for the reversal of neuromuscular blockade. Pharmacotherapy. 2007 Aug;27(8):1181-8. doi: 10.1592/phco.27.8.1181. PMID 17655516
- [Background] Chambers D, Paulden M, Paton F, Heirs M, Duffy S, Craig D, Hunter J, Wilson J, Sculpher M, Woolacott N. Sugammadex for the reversal of muscle relaxation in general anaesthesia: a systematic review and economic assessment. Health Technol Assess. 2010 Jul;14(39):1-211. doi: 10.3310/hta14390. PMID 20688009
- [Background] Sorgenfrei IF, Norrild K, Larsen PB, Stensballe J, Ostergaard D, Prins ME, Viby-Mogensen J. Reversal of rocuronium-induced neuromuscular block by the selective relaxant binding agent sugammadex: a dose-finding and safety study. Anesthesiology. 2006 Apr;104(4):667-74. doi: 10.1097/00000542-200604000-00009. PMID 16571960
- [Background] Sadleir PH, Russell T, Clarke RC, Maycock E, Platt PR. Intraoperative anaphylaxis to sugammadex and a protocol for intradermal skin testing. Anaesth Intensive Care. 2014 Jan;42(1):93-6. doi: 10.1177/0310057X1404200116. PMID 24471669
- [Background] Rahe-Meyer N, Fennema H, Schulman S, Klimscha W, Przemeck M, Blobner M, Wulf H, Speek M, McCrary Sisk C, Williams-Herman D, Woo T, Szegedi A. Effect of reversal of neuromuscular blockade with sugammadex versus usual care on bleeding risk in a randomized study of surgical patients. Anesthesiology. 2014 Nov;121(5):969-77. doi: 10.1097/ALN.0000000000000424. PMID 25208233

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients undergoing AVR, CABG or both were screened meeting preoperative inclusion criteria. Per the study design, elements of exclusion criteria incorporated intraoperative events. Patients were consented prior to the operation room with the understanding that they might be excluded depending on events in the operating room. Patients who screened and consented but did not participate in the study were not considered enrolled. A total of 90 participants were enrolled.
Period: Overall Study
Arm/Group | Sugammadex | Placebo
Started | 45 | 45
Completed | 40 | 43
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex | Placebo | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67.0 [62.0 to 72.0] | 66.0 [59.0 to 71.0] | 67.0 [60.0 to 71.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 37 | 40 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 44 | 45 | 89
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 41 | 41 | 82
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.39 (4.83) | 29.55 (4.61) | 29.47 (4.70)
Smoking [Count of Participants; unit: Participants]
  Current | 7 | 8 | 15
  Never | 21 | 19 | 40
  Prior | 17 | 18 | 35
Coexisting Medical Conditions [Count of Participants; unit: Participants]
  Hypertension | 37 | 32 | 69
  COPD | 1 | 1 | 2
  TIA/ Stroke | 2 | 1 | 3
HBA1c [Median (Inter-Quartile Range); unit: percentage of HbA1c] | 6.9 [6.3 to 7.4] | 6.2 [5.8 to 7.2] | 6.6 [5.9 to 7.3]
Preoperative Medications [Count of Participants; unit: Participants]
  Aspirin | 37 | 33 | 70
  Plavix | 2 | 2 | 4
  Angiotensin-converting enzyme inhibitors or Angiotensin II receptor blockers | 30 | 23 | 53
  Beta blockers | 33 | 23 | 56
  Statins | 40 | 31 | 71
  Other antihyperlipidemics | 7 | 5 | 12
ASA Class [Count of Participants; unit: Participants] — The American Society of Anesthesiologists (ASA) physical status classification system.
  ASA 1: A normal healthy patient. ASA 2: A patient with mild systemic disease. ASA 3: A patient with a severe systemic disease that is not life-threatening. ASA 4: A patient with a severe systemic disease that is a constant threat to life.
  ASA 5: A moribund patient who is not expected to survive without the operation.
  Class 1-3 were placed in a similar group as they were considered to have similar prognosis. Similarly Class 4-5 were considered to have worse prognosis.
  Participants
    </= 3 | 14 | 13 | 27
    4 or 5 | 31 | 32 | 63
STS Surgery Risk Score [Mean (Standard Deviation); unit: %] — The Society of Thoracic Surgeons (STS) score and other factors may be used to stratify patients into low, intermediate, and high risk . In general, an STS predicted risk of surgical mortality of 4%-8% is considered intermediate risk and 8% or greater is considered high risk.The STS score is based on age, gender, comorbidities (including hypertension, peripheral arterial disease, cerebrovascular disease, diabetes, and lung disease), and immediate preoperative condition (including presence of cardiogenic shock and whether the patient currently has heart failure).
  % | 1.58 (0.80) | 1.34 (.49) | 1.46 (0.68)
Type of Surgery [Count of Participants; unit: Participants]
  AVR | 5 | 8 | 13
  CABG | 34 | 34 | 68
  CABG plus AVR | 6 | 3 | 9
Surgical Factors: Characteristics [Count of Participants; unit: Participants]
  Redo sternotomy | 0 | 1 | 1
  Off Pump surgery | 1 | 0 | 1
Surgical Factors (Time) [Median (Inter-Quartile Range); unit: Minutes]
  Cardiopulmonary Bypass time | 89.2 [74.4 to 110.1] | 85.0 [68.8 to 95.2] | 86.0 [69.2 to 103.9]
  Cross clamp time | 68.7 [54.0 to 84.0] | 63.6 [54.2 to 78.9] | 66.0 [54.0 to 81.6]
RBCs (Units) [Count of Participants; unit: Participants]
  0 | 43 | 44 | 87
  1 | 1 | 1 | 2
  3 | 1 | 0 | 1
Platelets (units) [Count of Participants; unit: Participants]
  0 | 34 | 35 | 69
  1 | 11 | 10 | 21
FFP (units) [Count of Participants; unit: Participants]
  0 | 44 | 42 | 86
  1 | 1 | 1 | 2
  2 | 0 | 2 | 2
Intraoperative Tidal volume [Median (Inter-Quartile Range); unit: (ml/kg)] | 5.3 [4.3 to 6.5] | 5.7 [4.6 to 6.8] | 5.3 [4.3 to 6.8]
Pre-op Hemoglobin (g/dL) [Median (Inter-Quartile Range); unit: g/dL] | 13.9 [12.8 to 14.7] | 14.6 [13.6 to 15.3] | 14.2 [13.1 to 15.3]
Creatinine [Median (Inter-Quartile Range); unit: mg/dL] | 1.0 [.9 to 1.1] | .9 [.8 to 1.0] | 1 [.8 to 1.1]
Intraoperative opioids [Median (Inter-Quartile Range); unit: mcg]
  Total intraoperative Fentanyl | 400.0 [0 to 750.0] | 150.0 [0 to 750.0] | 250.0 [0 to 750.0]
  Total intraoperative Sufentanyl | 145.6 [0.0 to 370.4] | 250.5 [0.0 to 495.7] | 231.8 [0.0 to 426.0]
Intraoperative Fluids [Median (Inter-Quartile Range); unit: ml] — Note: patients that do not receive albumin can have a value of zero and therefore the mean or median can equal 0 as a result.
  ml
    Intraoperative crystalloids | 1950.0 [1400.0 to 2450.0] | 1900.0 [1400.0 to 2208.0] | 1900.0 [1400.0 to 2400.0]
    Intraoperative colloids | 0.0 [0.0 to 500.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 500.0]
PaO2/FiO2 ratio [Median (Inter-Quartile Range); unit: ratio] — PaO2/FiO2 ratio was assessed on first ABG in the ICU. It is the ratio of arterial oxygen partial pressure (PaO2 in mmHg) to fractional inspired oxygen (FiO2 ). Higher values are better.
  ratio | 224.6 [188.3 to 281.7] | 210.0 [180.0 to 276.7] | 220.0 [183.3 to 281.7]
Intraoperative Anesthetic: Rocuronium [Median (Inter-Quartile Range); unit: mg] | 150.0 [100.0 to 200.0] | 150.0 [100.0 to 200.0] | 150.0 [100.0 to 200.0]
Intraoperative Anesthetic: Midazolam [Median (Inter-Quartile Range); unit: mg] | 7.0 [5.0 to 8.0] | 7.0 [5.0 to 10.3] | 7.0 [5.0 to 9.9]
Intraoperative Anesthetic: Propofol [Median (Inter-Quartile Range); unit: mg] | 204.0 [120.0 to 501.0] | 185.0 [93.0 to 281.0] | 196.0 [108.0 to 455.0]

OUTCOME MEASURES:

1. Primary Outcome: Time to Extubation
Description: The primary outcome of this study aims to test the time to extubation among patients in the cardiothoracic ICU who have undergone isolated CABG.
Time Frame: Up to 2 weeks
Population: Of the 90 patients that were included in the study (45 in each group), a total of 68 patients underwent CABG, 13 AVR and 9 combined AVR and CABG.
Measure: Median (Inter-Quartile Range); unit: minutes
Groups:
- Sugammadex: Research pharmacy will provide the Sugammadex (2m/kg) vs. Placebo in a syringe.
  Sugammadex: The one time intravenous administration of the study and placebo compounds will be performed by CTICU nurses who will receive the drugs in a blinded fashion from the departmental research pharmacy.
- Placebo: Research pharmacy will provide the Sugammadex (2m/kg) vs. Placebo in a syringe.
  Placebo: The one time intravenous administration of the study and placebo compounds will be performed by CTICU nurses who will receive the drugs in a blinded fashion from the departmental research pharmacy.
Arm/Group | Sugammadex | Placebo
Number analyzed (Participants) | 45 | 45
minutes | 126.0 [84.0 to 274.0] | 219.0 [121.0 to 323.0]

2. Secondary Outcome: Negative Inspiratory Force
Description: NIF=Negative Inspiratory Force
Time Frame: Up to 2 weeks
Measure: Median (Inter-Quartile Range); unit: cm per H2O
Groups:
- Sugammadex Group: Sugammadex Group: Study Group
- Placebo Group: Placebo Group:Control Group
Arm/Group | Sugammadex Group | Placebo Group
Number analyzed (Participants) | 45 | 45
cm per H2O | -33.0 [-40.0 to -27.0] | -31.0 [-37 to -24]

3. Secondary Outcome: RSBI
Description: Rapid Shallow Breathing Index
Time Frame: Upto 2 weeks
Measure: Median (Inter-Quartile Range); unit: breaths/min/L
Groups:
- Sugammadex Group: Sugammadex Group:Study Group
- Placebo Group: Placebo Group: Control Group
Arm/Group | Sugammadex Group | Placebo Group
Number analyzed (Participants) | 45 | 45
breaths/min/L | 40.0 [28.9 to 60.6] | 32.7 [24.6 to 46.4]

4. Secondary Outcome: Length of ICU Stay
Description: Days in the ICU post opertaitvely
Time Frame: Up to 2 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Sugammadex Group | Placebo Group
Number analyzed (Participants) | 45 | 45
days | 2 [2 to 3] | 2 [2 to 3]

5. Secondary Outcome: Length of Hospital Stay
Description: Length of Hospital stay after surgery
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Sugammadex Group | Placebo Group
Number analyzed (Participants) | 45 | 45
Days | 5 [4 to 6] | 5 [4 to 6]

6. Secondary Outcome: New Dysrhythmia
Description: Any dysrhythmia after surgery in patients without history of dysrhythmia
Time Frame: Up to 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sugammadex Group | Placebo Group
Number analyzed (Participants) | 45 | 45
Participants | 3 | 6

7. Secondary Outcome: Change in Renal Function
Description: Change in renal function was defined as Creatinine elevation >0.5 mg/dl
Time Frame: Up to 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sugammadex Group | Placebo Group
Number analyzed (Participants) | 45 | 45
Participants | 5 | 3

8. Secondary Outcome: Postoperative CHF
Description: Postoperative congestive heart failure
Time Frame: Up to 2 weeks
Population: There was not statistically significant difference between the 2 groups. (p=1.0)
Measure: Count of Participants; unit: Participants
Arm/Group | Sugammadex Group | Placebo Group
Number analyzed (Participants) | 45 | 45
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were recorded during the hospitalization, an average of 5 days
Groups:
- Sugammadex: Patients received 2 mg/kg Sugammadex intravenously once in the postoperative period in a blinded fashion.
- Placebo: Patients received placebo intravenously once in the postoperative period in a blinded fashion.
Arm/Group | Sugammadex | Placebo
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 8/45 | 9/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex (N=45) | Placebo (N=45)
postoperative creatinine rise greater than 0.5 mg/dl (Renal and urinary disorders) | 5 (5) | 3 (3)
postoperative atrial fibrillation (Cardiac disorders) | 3 (3) | 6 (6)

LIMITATIONS AND CAVEATS:
First this was a single center study. Second, we excluded patients undergoing mitral valve surgeries or those with moderate to severe LV dysfunction, as these patients often have preexisting pulmonary edema. Third, seven patients in the study were randomized but did not receive study drug or placebo.These were analyzed as intention to treat. Extubation time was defined from study drug administration to extubation. This definition was different from our a priori planned protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT03196167/Prot_002.pdf
  • Statistical Analysis Plan (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT03196167/SAP_003.pdf
  • Informed Consent Form (2020-05-27): https://cdn.clinicaltrials.gov/large-docs/67/NCT03196167/ICF_001.pdf